CLINICAL TRIAL: NCT04418986
Title: Incisional Correction of Corneal Astigmatism During Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Collaborators: Baghdad Medical City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR200105
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: A randomized, parallel two-arm interventional study, the patients were divided into a 1:1 ratio, the study included eyes with visually significant cataract and preoperative corneal regular astigmatism between 0.75 and 2 Diopters undergoing phacoemulsification surgery. They were divided into two groups: controls underwent phacoemulsification with on-axis incision (CCI Group), and patients underwent phacoemulsification with opposite clear corneal incisions (OCCI Group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (CCI Group) (Sham Comparator): The Participants will undergo phacoemulsification with on-axis incision
  Interventions: Procedure: opposite clear corneal incisions (OCCI)
- Study (OCCI Group) (Active Comparator): The Participants will undergo phacoemulsification with opposite clear corneal incisions
  Interventions: Procedure: opposite clear corneal incisions (OCCI)

INTERVENTIONS:
Procedure: opposite clear corneal incisions (OCCI) — Coaxial small incision cataract surgery was performed for all cases using a 2.8 mm keratome placed at steep meridian and 1-mm paracentesis was made 90 degrees apart with a 20-gauge microvitrectomy blade. Surgery was performed with a 30-degree, 0.9-caliper phacoemulsification tip (microtip) with a divide and conquer technique.
  In the OCCI group, a single penetrating incision was created with 2.8 mm keratome in the clear cornea, 1.5 mm anterior to limbal blood vessels, centered over the steep meridian and opposite the phacoemulsification incision.

SUMMARY:
Today, cataract surgery is regarded as refractive surgery, mainly aiming emmetropia, and this makes eliminating corneal astigmatism is critical. Corneal astigmatism of more than 1 diopter has been reported in up to 45% of the cataract surgery candidates.

It is possible to reduce pre-existing corneal astigmatism by creating a clear corneal incision at the steep meridian of the cornea, however; creating a small incision can correct the only astigmatism up to 1 Diopter, and sometimes this method may not be easy to perform due to the location of steep meridian like the difficulty while creating a superonasal or inferonasal incision at the left eye. This approach is usually sufficient for correcting astigmatism less than 1 D in most eyes. An opposite side clear corneal incision (OCCI) could enhance the flattening effect on the cornea.

ELIGIBILITY:
Inclusion Criteria:

* Clear cornea
* No history of previous ocular surgery
* Central corneal thickness (CCT) <640

Exclusion Criteria:

* Irregular corneal astigmatism or lenticular astigmatism
* Corneal opacities or pathology like Fuch's endothelial dystrophy
* Previous ocular surgeries like glaucoma surgery or PKP or pterygium excision
* Posterior segment diseases and pathology
* Complicated phacoemulsification

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mean astigmatic correction | After 1 month of surgery
  Astigmatic correction change after the correction surgery
Mean surgically induced astigmatism | After 1 month of surgery
  Mean surgically induced astigmatism, measured by a vector-corrected method

SECONDARY OUTCOMES:
Change in visual acuity | After 1 month of surgery
  Uncorrected visual acuity and best corrected visual acuity after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ghazi al-Hariri Surgical Specialties Hospital, Baghdad, Bab-Almuadham, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code